CLINICAL TRIAL: NCT02724410
Title: Home Intravenous Versus Oral Antibiotics Following Appendectomy for Perforated Appendicitis in Children, a Randomized Controlled Trial
Brief Title: Role of Intravenous Versus Home Oral Antibiotics in Perforated Appendicitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-10-13B
Record Dates: First submitted 2016-03-15; First posted 2016-03-31 (Estimated); Results first posted 2022-03-23 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-02

CONDITIONS: Perforated Appendicitis
Keywords: appendectomy
MeSH Terms: conditions — Appendicitis | interventions — Ertapenem; Amoxicillin-Potassium Clavulanate Combination; Catheterization, Peripheral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- home intravenous ertapenem and PICC (Active Comparator): Placement of peripheral inserted central catheter (PICC) and completion of ten day antibiotic treatment with home (IV) ertapenem (Drug Class:carbapenem antibiotic) (15 mg/kg IV every twelve hours not to exceed 1 gm/day for ages <13; age 13 or greater, then 1 gm daily)
  Interventions: Drug: home intravenous ertapenem; Device: peripheral inserted central Catheter
- home oral amoxicillin-clavulanate (Experimental): Completion of ten day antibiotic treatment with home oral amoxicillin-clavulanate(Drug Class:beta lactam antibiotic)(15mg/kg every eight hours or 22.5mg/kg extended release tablets every twelve hours).
  Interventions: Drug: home oral amoxicillin-clavulanate

INTERVENTIONS:
Drug: home intravenous ertapenem — see arm description
  Other Names: Invanz
  Arms: home intravenous ertapenem and PICC
Drug: home oral amoxicillin-clavulanate — see arm description
  Other Names: Augmentin
  Arms: home oral amoxicillin-clavulanate
Device: peripheral inserted central Catheter — All patients undergoing home intravenous ertapenem will require placement of peripheral inserted central Catheter (PICC) for home delivery of antibiotics.
  Other Names: PICC
  Arms: home intravenous ertapenem and PICC

SUMMARY:
To compare the effect of a single-agent home intravenous (IV) versus oral antibiotic therapy on complication rates and resource utilization following appendectomy for perforated appendicitis

DETAILED DESCRIPTION:
Appendicitis is the most common cause of abdominal pain requiring emergent surgical intervention in children and approximately one third of patients present with perforation. Perforated appendicitis has been demonstrated to have a significant impact on patients and families due to the prolonged hospitalization, high complication rates, and tremendous economic burden from treatment. The most significant complication following operative treatment of perforated appendicitis is intra-abdominal abscess, which develops in approximately 20% of children following appendectomy in recent literature. Due to this frequent and morbid complication, continued research has been driven at determining the most efficacious and cost-effective postoperative antibiotic treatment regimen to reduce post-operative abscess. As postoperative abscess rates following appendectomy for perforated appendicitis remain high, the primary aim of this study was to evaluate a new postoperative antibiotic treatment regimen based on single daily dosing ertapenem while inpatient with randomization into ten day completion course of home antibiotics with IV ertapenem versus oral amoxicillin/clavulanate. The hypothesis is that the ertapenem based regimen will offer reduced rates of postoperative abscess, with no major difference between completion courses of home IV versus oral antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Patients 4-17 years of age with perforated acute appendicitis diagnosed at time of appendectomy.

Exclusion Criteria:

* Patients with a known severe allergy to penicillin (anaphylaxis), prior severe side effects from ertapenem or amoxicillin-clavulanate, pregnancy, or previous drainage procedure for abscess and/or fluid collection related to appendicitis.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2011-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brant T Heniford, M.D., Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Home Intravenous Ertapenem and PICC: Placement of peripheral inserted central catheter (PICC) and completion of ten day antibiotic treatment with home (IV) ertapenem (Drug Class: carbapenem antibiotic) (15 mg/kg IV every twelve hours not to exceed 1 gm/day for ages <13; age 13 or greater, then 1 gm daily)
  Peripheral inserted central Catheter: All patients undergoing home intravenous ertapenem will require placement of peripheral inserted central Catheter (PICC) for home delivery of antibiotics.
- Home Oral Amoxicillin-clavulanate: Completion of ten day antibiotic treatment with home oral amoxicillin-clavulanate (Drug Class: beta lactam antibiotic) (15mg/kg every eight hours or 22.5mg/kg extended release tablets every twelve hours).
Period: Overall Study
Arm/Group | Home Intravenous Ertapenem and PICC | Home Oral Amoxicillin-clavulanate
Started | 44 | 38
Completed | 44 | 38
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Home Intravenous Ertapenem and PICC | Home Oral Amoxicillin-clavulanate | Total
Number analyzed (Participants) | 44 | 38 | 82
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12.3 (3.6) | 10.1 (3.6) | 11.3 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 18 | 41
  Male | 21 | 20 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 24 | 19 | 43
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 15 | 17 | 32
Region of Enrollment [Number; unit: Participants]
  United States | 44 | 38 | 82
BMI [Mean (Standard Deviation); unit: kg/m^2] | 20.9 (5.8) | 17.9 (3.5) | 19.5 (5.0)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Postoperative Abscess
Description: Number of Postoperative Abscess, thirty-day postoperative
Time Frame: Thirty days after appendectomy
Measure: Count of Participants; unit: Participants
Arm/Group | Home Intravenous Ertapenem and PICC | Home Oral Amoxicillin-clavulanate
Number analyzed (Participants) | 44 | 38
Participants | 5 | 3
Statistical Analysis 1: Comparison: Home Intravenous Ertapenem and PICC vs Home Oral Amoxicillin-clavulanate; Test type: Other — Chi Square test of independence; p = 0.7188, Chi-squared

2. Primary Outcome: Number of Participants With Wound Infections
Description: Number of Wound Infections, 30-days postoperative
Time Frame: Thirty days following appendectomy
Measure: Count of Participants; unit: Participants
Arm/Group | Home Intravenous Ertapenem and PICC | Home Oral Amoxicillin-clavulanate
Number analyzed (Participants) | 44 | 38
Participants | 1 | 2
Statistical Analysis 1: Comparison: Home Intravenous Ertapenem and PICC vs Home Oral Amoxicillin-clavulanate; Test type: Other — Chi Square test of independence; p = .5933, Chi-squared

3. Primary Outcome: Number Participants With Readmission Within 30 Days
Description: Number of Readmission within 30 days postoperative
Time Frame: Thirty days following appendectomy
Measure: Count of Participants; unit: Participants
Arm/Group | Home Intravenous Ertapenem and PICC | Home Oral Amoxicillin-clavulanate
Number analyzed (Participants) | 44 | 38
Participants | 6 | 6
Statistical Analysis 1: Comparison: Home Intravenous Ertapenem and PICC vs Home Oral Amoxicillin-clavulanate; Test type: Other — Chi Square test of independence; p > .99, Chi-squared

4. Primary Outcome: Hospital Charge
Description: Cost of Hospital services
Time Frame: Thirty days following appendectomy
Measure: Mean (Standard Deviation); unit: Dollars
Arm/Group | Home Intravenous Ertapenem and PICC | Home Oral Amoxicillin-clavulanate
Number analyzed (Participants) | 37 | 31
Dollars | 47564.3 (9057.59) | 34227.79 (8104.65)
Statistical Analysis 1: Comparison: Home Intravenous Ertapenem and PICC vs Home Oral Amoxicillin-clavulanate; Test type: Other — T-test for difference between groups; p < .0001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Home Intravenous Ertapenem and PICC | Home Oral Amoxicillin-clavulanate
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/44 | 2/38
Other Adverse Events (participants affected / at risk) | 0/44 | 0/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Home Intravenous Ertapenem and PICC (N=44) | Home Oral Amoxicillin-clavulanate (N=38)
Adinamic ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No